CLINICAL TRIAL: NCT04863495
Title: A Multi-Center Observational Study of Couples Across the Trajectory of Dementia
Brief Title: Couples Lived Experience
Status: Active, not recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-01966
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease; Dementia of Alzheimer Type
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a longitudinal study with regular quantitative assessments of all participants every six months for 3 years. The quantitative portion of the study will recruit couples, consisting of individuals over the age of 65 who are in a committed relationship. Both members of the couple must be willing to participate at baseline. The assessment is in two parts. In the first part, each member of the couple will be asked the following: demographic information, mental health history, self-reported physical and emotional health, measures of emotional and mental health, personality, relationship and attachment style, social support and self-efficacy. Then each member of the study couple will be asked a series of questions to determine whether they consider themselves a caregiver. If they do, individuals will be asked to respond to additional caregiver questionnaires. Follow-ups will occur every six months for the study couples for a total of three years from the baseline visit. Each visit, the entire assessment except for demographic questions, will be re-administered to each individual in the couple. At the end of each questionnaire battery, individuals will be screened for cognitive impairment and those who are in the middle to advanced stages of dementia will no longer participate. Recruitment will end when 600 individuals (300 couples,150 couples at each site) are enrolled in the longitudinal portion of the study. All study visits will be conducted virtually via Zoom or WebEx video conferencing. Analyses will be conducted to determine the association between changes in dyadic relationship and changes in mental health and cognitive outcomes, to elucidate how relationship characteristics impact health and well-being as perceived by each member of the dyad.

ELIGIBILITY:
Longitudinal Portion

Inclusion Criteria:

1. Community dwelling older adult aged 65 years or older
2. Must speak English as the study measures are not validated in other languages.
3. Must express intent to commit to ongoing participation in longitudinal study with assessments every 6 months for 3 years,
4. Is part of a couple and their spouse/partner is also willing to participate in the project. All couples, regardless of sexual orientation or gender preference are eligible to participate
5. Both members of the couple must cohabitate at the time of enrollment.
6. Must have stable internet connection and capability to stream video with audio.
7. A subset of the longitudinal study participants (selected at random) will be invited to be participate in a focus group upon completion of the last (3 year) quantitative assessment. These participants must be willing to have their comments recorded.

Exclusion Criteria:

1. Any individual with a prior diagnosis of schizophrenia or other psychotic disorder.
2. Individual is unable to complete the informed consent process
3. Any individual with a prior diagnosis of a chronic disabling medical condition that would make it impossible to participate in a focus group via Zoom or WebEx.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: All genders, over the age of 65 that are community dwelling and in a committed relationship with an individual (also over the age of 65) that also agrees to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-04-19 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Score on Geriatric Depression Scale (GDS-15) | Day 0
  This is a 15-item self-report measure of symptoms of depression among older adults. It consists of 15 questions in which participants are asked to respond by answering either 'yes' or 'no' in reference to how they felt over the past week. For each question, dependent on the answer, 1 point is given. Total range of score is 0-15. A score > 5 points is suggestive of depression. A score ≥ 10 points is almost always indicative of depression. A score > 5 points should warrant a follow-up comprehensive assessment.
Score on Geriatric Depression Scale (GDS-15) | Month 6
  This is a 15-item self-report measure of symptoms of depression among older adults. It consists of 15 questions in which participants are asked to respond by answering either 'yes' or 'no' in reference to how they felt over the past week. For each question, dependent on the answer, 1 point is given. Total range of score is 0-15. A score > 5 points is suggestive of depression. A score ≥ 10 points is almost always indicative of depression. A score > 5 points should warrant a follow-up comprehensive assessment.
Score on Geriatric Depression Scale (GDS-15) | Month 12
  This is a 15-item self-report measure of symptoms of depression among older adults. It consists of 15 questions in which participants are asked to respond by answering either 'yes' or 'no' in reference to how they felt over the past week. For each question, dependent on the answer, 1 point is given. Total range of score is 0-15. A score > 5 points is suggestive of depression. A score ≥ 10 points is almost always indicative of depression. A score > 5 points should warrant a follow-up comprehensive assessment.
Score on Geriatric Depression Scale (GDS-15) | Month 18
  This is a 15-item self-report measure of symptoms of depression among older adults. It consists of 15 questions in which participants are asked to respond by answering either 'yes' or 'no' in reference to how they felt over the past week. For each question, dependent on the answer, 1 point is given. Total range of score is 0-15. A score > 5 points is suggestive of depression. A score ≥ 10 points is almost always indicative of depression. A score > 5 points should warrant a follow-up comprehensive assessment.
Score on Geriatric Depression Scale (GDS-15) | Month 24
  This is a 15-item self-report measure of symptoms of depression among older adults. It consists of 15 questions in which participants are asked to respond by answering either 'yes' or 'no' in reference to how they felt over the past week. For each question, dependent on the answer, 1 point is given. Total range of score is 0-15. A score > 5 points is suggestive of depression. A score ≥ 10 points is almost always indicative of depression. A score > 5 points should warrant a follow-up comprehensive assessment.
Score on Geriatric Depression Scale (GDS-15) | Month 30
  This is a 15-item self-report measure of symptoms of depression among older adults. It consists of 15 questions in which participants are asked to respond by answering either 'yes' or 'no' in reference to how they felt over the past week. For each question, dependent on the answer, 1 point is given. Total range of score is 0-15. A score > 5 points is suggestive of depression. A score ≥ 10 points is almost always indicative of depression. A score > 5 points should warrant a follow-up comprehensive assessment.
Score on Geriatric Depression Scale (GDS-15) | Month 36
  This is a 15-item self-report measure of symptoms of depression among older adults. It consists of 15 questions in which participants are asked to respond by answering either 'yes' or 'no' in reference to how they felt over the past week. For each question, dependent on the answer, 1 point is given. Total range of score is 0-15. A score > 5 points is suggestive of depression. A score ≥ 10 points is almost always indicative of depression. A score > 5 points should warrant a follow-up comprehensive assessment.
Score on Beck Anxiety Inventory (BAI) Report | Day 0
  This is a 21-item self-report measure of symptoms of anxiety, including experiences of physical symptoms associated with anxiety. Participants are asked to rate how each symptom bothered them during the past month, on a 4-point scale from 0 ("Not at all") to 3 ("Severely-it bothered me a lot"). The total range of score is 0-63. The higher the score the higher the severity of symptoms.
Score on Beck Anxiety Inventory (BAI) Report | Month 6
  This is a 21-item self-report measure of symptoms of anxiety, including experiences of physical symptoms associated with anxiety. Participants are asked to rate how each symptom bothered them during the past month, on a 4-point scale from 0 ("Not at all") to 3 ("Severely-it bothered me a lot"). The total range of score is 0-63. The higher the score the higher the severity of symptoms.
Score on Beck Anxiety Inventory (BAI) Report | Month 12
  This is a 21-item self-report measure of symptoms of anxiety, including experiences of physical symptoms associated with anxiety. Participants are asked to rate how each symptom bothered them during the past month, on a 4-point scale from 0 ("Not at all") to 3 ("Severely-it bothered me a lot"). The total range of score is 0-63. The higher the score the higher the severity of symptoms.
Score on Beck Anxiety Inventory (BAI) Report | Month 18
  This is a 21-item self-report measure of symptoms of anxiety, including experiences of physical symptoms associated with anxiety. Participants are asked to rate how each symptom bothered them during the past month, on a 4-point scale from 0 ("Not at all") to 3 ("Severely-it bothered me a lot"). The total range of score is 0-63. The higher the score the higher the severity of symptoms.
Score on Beck Anxiety Inventory (BAI) Report | Month 24
  This is a 21-item self-report measure of symptoms of anxiety, including experiences of physical symptoms associated with anxiety. Participants are asked to rate how each symptom bothered them during the past month, on a 4-point scale from 0 ("Not at all") to 3 ("Severely-it bothered me a lot"). The total range of score is 0-63. The higher the score the higher the severity of symptoms.
Score on Beck Anxiety Inventory (BAI) Report | Month 30
  This is a 21-item self-report measure of symptoms of anxiety, including experiences of physical symptoms associated with anxiety. Participants are asked to rate how each symptom bothered them during the past month, on a 4-point scale from 0 ("Not at all") to 3 ("Severely-it bothered me a lot"). The total range of score is 0-63. The higher the score the higher the severity of symptoms.
Score on Beck Anxiety Inventory (BAI) Report | Month 36
  This is a 21-item self-report measure of symptoms of anxiety, including experiences of physical symptoms associated with anxiety. Participants are asked to rate how each symptom bothered them during the past month, on a 4-point scale from 0 ("Not at all") to 3 ("Severely-it bothered me a lot"). The total range of score is 0-63. The higher the score the higher the severity of symptoms.
Score on Physical Health Questionnaire | Day 0
  Three questions to assess subjective evaluation of their own health: (1) How would you rate your overall physical health at the present time? (On a 4-point scale from 4 (poor) to 1 (excellent)); (2) Is your health now better, about the same or worse than it was five years ago? (On a 3-point scale; 3 (worse), 2 (about the same), 1 (better)); and (3) How much do your physical health troubles stand in the way of your doing the things you want to do? (On a 3-point scale; 3 (a great deal); 2 (a little (some)); 1 (not at all)). The sum of the 3 questions is used to measure SRH. Possible scores ranged from 3 (least healthy) to 10 (healthiest).
Score on Physical Health Questionnaire | Month 6
  Three questions to assess subjective evaluation of their own health: (1) How would you rate your overall physical health at the present time? (On a 4-point scale from 4 (poor) to 1 (excellent)); (2) Is your health now better, about the same or worse than it was five years ago? (On a 3-point scale; 3 (worse), 2 (about the same), 1 (better)); and (3) How much do your physical health troubles stand in the way of your doing the things you want to do? (On a 3-point scale; 3 (a great deal); 2 (a little (some)); 1 (not at all)). The sum of the 3 questions is used to measure SRH. Possible scores ranged from 3 (least healthy) to 10 (healthiest).
Score on Physical Health Questionnaire | Month 12
  Three questions to assess subjective evaluation of their own health: (1) How would you rate your overall physical health at the present time? (On a 4-point scale from 4 (poor) to 1 (excellent)); (2) Is your health now better, about the same or worse than it was five years ago? (On a 3-point scale; 3 (worse), 2 (about the same), 1 (better)); and (3) How much do your physical health troubles stand in the way of your doing the things you want to do? (On a 3-point scale; 3 (a great deal); 2 (a little (some)); 1 (not at all)). The sum of the 3 questions is used to measure SRH. Possible scores ranged from 3 (least healthy) to 10 (healthiest).
Score on Physical Health Questionnaire | Month 18
  Three questions to assess subjective evaluation of their own health: (1) How would you rate your overall physical health at the present time? (On a 4-point scale from 4 (poor) to 1 (excellent)); (2) Is your health now better, about the same or worse than it was five years ago? (On a 3-point scale; 3 (worse), 2 (about the same), 1 (better)); and (3) How much do your physical health troubles stand in the way of your doing the things you want to do? (On a 3-point scale; 3 (a great deal); 2 (a little (some)); 1 (not at all)). The sum of the 3 questions is used to measure SRH. Possible scores ranged from 3 (least healthy) to 10 (healthiest).
Score on Physical Health Questionnaire | Month 24
  Three questions to assess subjective evaluation of their own health: (1) How would you rate your overall physical health at the present time? (On a 4-point scale from 4 (poor) to 1 (excellent)); (2) Is your health now better, about the same or worse than it was five years ago? (On a 3-point scale; 3 (worse), 2 (about the same), 1 (better)); and (3) How much do your physical health troubles stand in the way of your doing the things you want to do? (On a 3-point scale; 3 (a great deal); 2 (a little (some)); 1 (not at all)). The sum of the 3 questions is used to measure SRH. Possible scores ranged from 3 (least healthy) to 10 (healthiest).
Score on Physical Health Questionnaire | Month 30
  Three questions to assess subjective evaluation of their own health: (1) How would you rate your overall physical health at the present time? (On a 4-point scale from 4 (poor) to 1 (excellent)); (2) Is your health now better, about the same or worse than it was five years ago? (On a 3-point scale; 3 (worse), 2 (about the same), 1 (better)); and (3) How much do your physical health troubles stand in the way of your doing the things you want to do? (On a 3-point scale; 3 (a great deal); 2 (a little (some)); 1 (not at all)). The sum of the 3 questions is used to measure SRH. Possible scores ranged from 3 (least healthy) to 10 (healthiest).
Score on Physical Health Questionnaire | Month 36
  Three questions to assess subjective evaluation of their own health: (1) How would you rate your overall physical health at the present time? (On a 4-point scale from 4 (poor) to 1 (excellent)); (2) Is your health now better, about the same or worse than it was five years ago? (On a 3-point scale; 3 (worse), 2 (about the same), 1 (better)); and (3) How much do your physical health troubles stand in the way of your doing the things you want to do? (On a 3-point scale; 3 (a great deal); 2 (a little (some)); 1 (not at all)). The sum of the 3 questions is used to measure SRH. Possible scores ranged from 3 (least healthy) to 10 (healthiest).
Score on EuroQol Questionnaire Global quality of life | Day 0
  This scale assesses the respondent's overall quality of life. The respondent is asked to rate how good or bad his overall quality of life is on the day of administration on a scale of 0-100 with 100 being "best imaginable quality of life" and 0 being the "worst imaginable quality of life"
Score on EuroQol Questionnaire Global quality of life | Month 6
  This scale assesses the respondent's overall quality of life. The respondent is asked to rate how good or bad his overall quality of life is on the day of administration on a scale of 0-100 with 100 being "best imaginable quality of life" and 0 being the "worst imaginable quality of life"
Score on EuroQol Questionnaire Global quality of life | Month 12
  This scale assesses the respondent's overall quality of life. The respondent is asked to rate how good or bad his overall quality of life is on the day of administration on a scale of 0-100 with 100 being "best imaginable quality of life" and 0 being the "worst imaginable quality of life"
Score on EuroQol Questionnaire Global quality of life | Month 18
  This scale assesses the respondent's overall quality of life. The respondent is asked to rate how good or bad his overall quality of life is on the day of administration on a scale of 0-100 with 100 being "best imaginable quality of life" and 0 being the "worst imaginable quality of life"
Score on EuroQol Questionnaire Global quality of life | Month 24
  This scale assesses the respondent's overall quality of life. The respondent is asked to rate how good or bad his overall quality of life is on the day of administration on a scale of 0-100 with 100 being "best imaginable quality of life" and 0 being the "worst imaginable quality of life"
Score on EuroQol Questionnaire Global quality of life | Month 30
  This scale assesses the respondent's overall quality of life. The respondent is asked to rate how good or bad his overall quality of life is on the day of administration on a scale of 0-100 with 100 being "best imaginable quality of life" and 0 being the "worst imaginable quality of life"
Score on EuroQol Questionnaire Global quality of life | Month 36
  This scale assesses the respondent's overall quality of life. The respondent is asked to rate how good or bad his overall quality of life is on the day of administration on a scale of 0-100 with 100 being "best imaginable quality of life" and 0 being the "worst imaginable quality of life"
Number of participants with status change | Month 36
  Status changes include but are not limited to residential care placement, move to live with another relative, death

CONTACTS AND LOCATIONS:
Overall Officials: Mary Mittelman, DrPH, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - Boston University, Bedford, Massachusetts
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Mary.Mittelman@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Mittelman MS, O'Connor MK, Donley T, Epstein-Smith C, Nguyen A, Nicholson R, Salant R, Shirk SD, Stevenson E. Longitudinal study: understanding the lived experience of couples across the trajectory of dementia. BMC Geriatr. 2021 Oct 15;21(1):558. doi: 10.1186/s12877-021-02503-4. PMID 34654375